CLINICAL TRIAL: NCT04831463
Title: The Effect of Increasising Health Awareness Program on Health Perceptıons and Responsıbılıtıes of Immıgrant Men (IHAP) on Perceived Stress Levels, Attitudes Towards Utiling Healthcare Services and Coping Strategies
Brief Title: The Effect of the Program on the Health Perceptions and Responsibilities of Immigrant Men on Utiling Healthcare Services
Acronym: IHAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilknur Aydin Avci, Head of Nursing Department, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-91
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Health Care Utilization; Men
Keywords: Immigrant Health, Men's Health, Health Promotion
MeSH Terms: conditions — Patient Acceptance of Health Care; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental (N = 49) received a short-term IHAPIM program by one-on-one interview (5 week, 1 hr per week, 10 hr in total).
  Interventions: Behavioral: Increasising Health Awareness Program for Immigrant Men
- control group (No Intervention): Firstly, Pre-tests were applied to the men in the control group. No intervention was applied to this group. Post-tests were made 3 months after finished intervention which applied to experimental group.

INTERVENTIONS:
Behavioral: Increasising Health Awareness Program for Immigrant Men — The IHAPIM program is a health promotion intervention. The aim of intervention improve health perception and responsibilitiy
  Arms: experimental group

SUMMARY:
Aims The study aims to examine the effect of "IHAPIM" program on health perceptions, health responsibilities, perceived stress level, attitudes towards utiling health care services and the types of coping strategies of immigrant men.

Design This study is a two centre, double-blind, randomized controlled trial. Methods We attempt to report this randomized controlled trial to comply with the SPIRIT. The study population consist of 95 immigrant men live at north of Turkey. The study, between March 2020-March 2021 were held in the two district predominantly immigrants. The participants were randomly divided into experimental and control group. The experimental (N = 49) received a short-term IHAPIM program (5 week, 1 hr per week, 10 hr in total). Measurements were obtained during pre- and post-test from experimental and control group (N = 46). In this study, participants and statistician who conducted the research blinded.

Discussion The efficacy of health promotion interventions are known. However, the health promotion interventions for immigrants men performed by public health nurse are not available. At the same time, the effect of health promotion interventions for immigrants men are unknown.

Impact This study is expected to provide a piece of credible evidence of the the health promotion interventions for immigrants men performed by public health nurse and efficacy of health perceptions, health responsibilities, perceived stress level, attitudes towards utiling health care services and the types of coping strategies in immigrant men group. It is assumed that health promotion interventions specific to male health and sensitive to the language of immigrants lead to a beneficial results on health perceptions, health responsibilities, perceived stress level, attitudes towards utiling health care services and the types of coping strategies in immigrant men. If "IHAPIM" program perform in practice by public heath nurse. It can be effectively improve immigrant men's health variables such as health perceptions, health responsibilities, perceived stress level, attitudes towards utiling health care services and the types of coping strategies.

DETAILED DESCRIPTION:
This study was carried out in order to examine the effect of the "Increasising Health Awareness Program for Immigrant Men " (IHAPIM), which was prepared based on the Transition Theory of Meleis, on the health perceptions, health responsibilities, perceived stress levels, attitudes towards utiling health care services and the types of coping strategies of immigrant men.

This study, which was planned in accordance with the principles of a randomized controlled double-blind pre-test post-test control group experimental study, was conducted with immigrant males between the ages of 18 and 50, living in Canik and İlkadım districts of Samsun, where immigrants live mainly. The randomized clinical trial was based on the guidelines proposed by the SPIRIT 2013 Statement. The data of the study were collected in Samsun / Ilkadım and Canık District between May 2020 and November 2020. Randomization an experimental group and a control group formed using the research randomizer software. the program used random numbers to select participants and randomly assign them to the experimental or control group (total 95 immigrant men). In this study, immigrant men do not know that they are in the experimental or control group, and the statistician who conducted the research does not know which data belong to which group. Blinding is done in this way. The study was completed with 49 men in the experimental group and 46 men in the control group. The experimental (N = 49) received a short-term IHAPIM program by one-on-one interview (5 week, 1 hr per week). The data of the study were collected using personal information form, health perception scale, health responsibility sub-dimension of healthy lifestyle behaviors scale, perceived stress scale, stress coping methods scale and the scale of determining the attitudes of immigrants towards using health services.

personal information form; the form was developed by the researcher and consists of questions involving sociodemographic characteristics (age, marital status, education status, etc.) health perception scale; Health perceptions of immigrant men were evaluated with a visual number scale. There is a question on the scale. Information on how to fill the scale as parentheses information at the end of the question scored between 1-10, which is easy to understand, which immigrant men can answer on their own ('0' on this scale indicates that you evaluate your questioned situation very badly, the increase of the score is improving your assessment of your questioned situation, and the '10' score is shows that your assessment of your situation is very good).

health responsibility sub-dimension of healthy lifestyle behaviors scale; In measuring the level of responsibility for an individual's health, the healthy lifestyle behaviors scale, which was developed by Walker, Sechrist and Pender in 1987 and adapted to Arabic in 1998 by Hadad et al. is the scale that determines the extent to which they participate in health. All items of the healthy lifestyle behaviors scale are positive. There is no reverse matter. Marking is done on 4 Likert type scales. A score of 1 is given for an answer "Never", 2 points for an answer "Sometimes", 3 points for an answer "Often" and 4 points for an answer "Regularly". Health responsibility sub-dimension of healthy lifestyle behaviors scale 2, 7, 15,20,28,31,33,42,43,46. It consisted of a total of 10 items including items. The lowest score is 10, the highest score is 40. The reliability coefficients of the scale are α 0.90.

perceived stress scale; The Perceived Stress Scale, developed by Cohen, Kamarc and Mermelstein (1983), is the most commonly used tool of this type. Chaaya et al. In 2010, its validity and reliability in Arabic was made. The scale consists of 10 items. It was developed to evaluate to what extent the individual perceived his life as unpredictable, uncontrollable or overloaded in the last month. The scale is in the 5-point Likert type (1- never, 2- almost never, 3- sometimes, 4- often 5- very often), and its four items are reverse (4th, 5th, 7th, 8th items), six of its articles are plainly worded (1st, 2nd, 3rd, 6th, 9th, 10th items). The lowest score that can be obtained from the scale is 0, and the highest score is 40. The scale is evaluated over the total score, and the higher the scores indicate that the stress is perceived high. The Arabic reliability coefficients of the scale are α 0.87.

types of coping strategies; The study of the "Ways of Coping Inventory" scale developed by Folkman and Lazarus (1980) in order to determine the ways individuals use to deal with general or significant stress situations, the Arabic validity and reliability was conducted by Alghamdi (2020). The "Coping with Stress Scale" consists of two groups, 14 sub-dimensions and 28 items, as compatible and incompatible. Harmonious coping methods; active coping, positive reframing, planning, acceptance, religion, humor, using emotional social support support), using useful social support (using instrumental support), incompatible coping methods; behavioral disengagement, denial, substance use, focusing on the problem and venting, mental self-distraction, self-blame. The Likert-type scale scored between 1 and 4 does not have a total score. Arabic validity and reliability study of the scale was conducted in 2018 and the reliability coefficient was found to be α 0.80 in the Arabic version of the scale.

the scale of determining the attitudes towards utiling health care services; Developed in Arabic by Avci and Korkmaz in 2019 in order to determine the attitudes of immigrants towards using health services, the scale for determining the attitudes of immigrants towards using health services consists of 26 items. The scale consists of 4 sub-dimensions: health awareness, factors affecting admission to health services, delivery of health services, and access to health services. Answers given to each statement in the scale are in 5-point Likert type and all statements are positive. Scores obtained from sub-dimensions: between 4-20 points for health awareness sub-dimension; Between 4-20 points for the factors affecting the application to health services sub-dimension; It ranges between 5-25 points for the sub-dimension of the way health services are provided and 5-25 points for the sub-dimension of access to health services. The total scores obtained from the scale range from 18 to 90 points. The fact that the scores obtained from the scale subscale and the total score are high indicates that the immigrants have a good attitude towards using health services. Cronbach's alphas in the validity and reliability study of the scale are as follows: Cronbach's Alpha reliability coefficient of the health awareness sub-dimension (0.63), the Cronbach's Alpha reliability coefficient (0.73) of the factors affecting admission to health services, the Cronbach's Alpha reliability coefficient of the sub-dimension of how health services are provided (0.60), and Cronbach's Alpha reliability coefficient of access to health services sub-dimension is (0.71). The total Cronbach's alpha reliability coefficient of the scale for determining the attitudes of immigrants towards using health services is 0.72.

Evaluation of Data SPSS 23.0 statistical package program (Statistical Package for the Social Sciences, Chicago, Illinois) was used for statistical analysis and evaluation of the data. Whether the data showed normal distribution was checked with the Kolmogorov-Smirnov test. Mann Whitney U test were used to compare data between groups according to normality test. Wilcoxon test were used to compare the pre-test and post-test values within the group. The Chi-square test and two ratio tests were used to analyze categorical data. Significance level was taken as p <0.05.

Funding: Financial support of the research provided by the Project Management Office of Ondokuz Mayis University. PYO.SBF.1904.20.002.

Ethical aspects: Study approval was given by Ondokuz Mayıs University Ethıcs Commıttee For Socıal And Humanıtıes Research. (Decision No: 2019-91). All participants were informed about tis study and obtained orat-written informed consents.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Be between the ages of 18 and 50
* Being a male
* No communication barriers
* Being a immigrant
* To be able to read and write Arabic language

Exclusion Criteria:

* Being younger than 18 or over 50
* Be woman
* Inability to communicate with any problem such as hearing problem, speech impediment
* Living undocumented
* Refusing to participate in the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The utiling of healthcare services by immigrant men is lower than immigrant women. Only men were recruited.
Enrollment: 100 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Increasing health perception and responsibility of immigrant men | 3 month
  After health promotion intervention (IHAPIM) this outcome will obtained

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Aydin AVCI, Prof., Study Director — Ondokuz Mayıs University; Metin Yılmaz, Prof., Study Chair — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)